CLINICAL TRIAL: NCT03016871
Title: A Phase II Trial of Response-Adapted Second-Line Therapy for Hodgkin Lymphoma Using Anti-PD-1 Antibody Nivolumab ? ICE Chemotherapy as a Bridge to Autologous Hematopoietic Cell Transplant (NICE Trial)
Brief Title: Nivolumab, Ifosfamide, Carboplatin, and Etoposide as Second-Line Therapy in Treating Patients With Refractory or Relapsed HL
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 16403; NCI-2016-02038 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 16403 (Other: City of Hope Medical Center)
Record Dates: First submitted 2017-01-06; First posted 2017-01-11 (Estimated); Results first posted 2024-10-09 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Recurrent Hodgkin Lymphoma; Refractory Hodgkin Lymphoma
MeSH Terms: conditions — Hodgkin Disease | interventions — Carboplatin; Etoposide; Ifosfamide; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A (nivolumab, etoposide, ifosfamide, carboplatin) (Experimental): Patients receive nivolumab IV over 30 minutes on day 1. Cycles repeat every 14 days for 6 weeks in the absence of disease progression or unacceptable toxicity. Patients with CR or PR receive nivolumab for an additional 6 weeks. Patients with only SD after 6-week nivolumab treatment receive nivolumab for an additional 6 weeks or receive nivolumab IV over 30 minutes on day 1, etoposide IV on days 1-3, ifosfamide IV continuously over 24 hours on day 2, and carboplatin IV on day 2 every 21 days for 6 weeks per physician/investigator's discretion. Patients with PD after 6-week nivolumab treatment or patients with PR, SD, or PD after 12-week nivolumab treatment receive nivolumab IV over 30 minutes on day 1, etoposide IV on days 1-3, ifosfamide IV continuously over 24 hours on day 2, and carboplatin IV on day 2. Treatment repeats every 21 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Carboplatin; Drug: Etoposide; Drug: Ifosfamide; Other: Laboratory Biomarker Analysis; Biological: Nivolumab
- Cohort B (nivolumab, etoposide, ifosfamide, carboplatin) (Experimental): Patients receive nivolumab IV over 30 minutes on cycle 1 (cycle 1 is 14 days), day 1 in the absence of disease progression or unacceptable toxicity. Beginning in cycle 2, patients receive nivolumab IV over 30 minutes on day 1, etoposide IV on days 1-3, ifosfamide IV continuously over 24 hours on day 2, and carboplatin IV on day 2. Treatment repeats every 21 days for up to 3 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Carboplatin; Drug: Etoposide; Drug: Ifosfamide; Other: Laboratory Biomarker Analysis; Biological: Nivolumab

INTERVENTIONS:
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16; VP 16-213; VP-16; VP-16-213; VP16
Drug: Ifosfamide — Given IV
  Other Names: Asta Z 4942; Asta Z-4942; Cyfos; Holoxan; Holoxane; Ifex; IFO; IFO-Cell; Ifolem; Ifomida; Ifomide; Ifosfamidum; Ifoxan; IFX; Iphosphamid; Iphosphamide; Iso-Endoxan; Isoendoxan; Isophosphamide; Mitoxana; MJF 9325; MJF-9325; Naxamide; Seromida; Tronoxal; Z 4942; Z-4942
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo

SUMMARY:
This phase II trial studies the side effects of nivolumab and to see how well it works when given together with ifosfamide, carboplatin, and etoposide in treating patients with Hodgkin lymphoma that has come back (relapsed) and does not respond to treatment (refractory). Immunotherapy with monoclonal antibodies such as nivolumab, may help the body?s immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Drugs used in chemotherapy, such as ifosfamide, carboplatin and etoposide, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving nivolumab, ifosfamide, carboplatin and etoposide may work better in treating patients with Hodgkin lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the anti-tumor activity of nivolumab as single agent and in combination with ifosfamide, carboplatin, etoposide (ICE) chemotherapy (nivolumab [N]ICE) as assessed by complete response (CR) rate prior to autologous hematopoietic cell transplantation.

II. To estimate the proportion of patients experiencing unacceptable adverse events. (Cohort B) III. To assess the safety and tolerability of nivolumab + ICE chemotherapy through evaluation of toxicities, including type, frequency, severity, attribution, time course, and duration. (Cohort B) IV. To obtain estimate of overall response rate (ORR), complete response rate, response duration and survival (overall and event-free). (Cohort B) V. Summarize stem cell mobilization outcomes (e.g., total CD34+ cell yield, number of apheresis days, proportion of patients who achieve >= 2 x 10^6 CD34+ cells/kg). (Cohort B) VI. Evaluate Hodgkin lymphoma biological markers in subjects treated with nivolumab. (Cohort B)

SECONDARY OBJECTIVES:

I. Assess the safety and tolerability of nivolumab +/- ICE chemotherapy through evaluation of toxicities, including type, frequency, severity, attribution, time course and duration.

II. Obtain estimates of overall response rate (ORR), response duration and survival (overall and event-free).

III. Summarize stem cell mobilization outcomes (e.g., total CD34+ cell yield, number of apheresis days, proportion of patients who achieve >= 2 x 10^6 CD34+ cells/kg).

IV. Evaluate Hodgkin lymphoma biological markers in subjects treated with nivolumab.

V. Among subjects who undergo autologous hematopoietic cell transplantation (AHCT), estimate the post-AHCT overall/progression free survival (PFS) probability and cumulative incidence of relapse/progression, non-relapse mortality (NRM) at 100-days, 1-year and 2-years.

VI. Among subjects who undergo autologous hematopoietic cell transplantation (AHCT), characterize post-AHCT toxicities during the first 30- and 100- days post stem cell infusion by type, frequency, severity, attribution, time course and duration.

VII. Among subjects who undergo autologous hematopoietic cell transplantation (AHCT), evaluate short and long-term post-AHCT complications, including: delayed engraftment (neutrophil and platelet) and infection, graft versus host disease and sinusoidal obstruction syndrome.

EXPLORATORY OBJECTIVES:

I. Collect deoxyribonucleic acid (DNA)/ribonucleic acid (RNA) from lymphoma specimens and serial plasma samples for future biomarker evaluation.

II. Evaluate potential changes in Hodgkin lymphoma biological markers of patients treated with nivolumab.

OUTLINE: Patients are sequentially assigned to 1 of 2 cohorts.

COHORT A: Patients receive nivolumab intravenously (IV) over 30 minutes on day 1. Cycles repeat every 14 days for 6 weeks in the absence of disease progression or unacceptable toxicity. Patients with CR or partial response (PR) receive nivolumab for an additional 6 weeks. Patients with only stable disease (SD) after 6-week nivolumab treatment receive nivolumab for an additional 6 weeks or receive nivolumab IV over 30 minutes on day 1, etoposide IV on days 1-3, ifosfamide IV continuously over 24 hours on day 2, and carboplatin IV on day 2 every 21 days for 6 weeks per physician/investigator's discretion. Patients with progressive disease (PD) after 6-week nivolumab treatment or patients with PR, SD, or PD after 12-week nivolumab treatment receive nivolumab IV over 30 minutes on day 1, etoposide IV on days 1-3, ifosfamide IV continuously over 24 hours on day 2, and carboplatin IV on day 2. Treatment repeats every 21 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity.

COHORT B: Patients receive nivolumab IV over 30 minutes on cycle 1 (cycle 1 is 14 days), day 1 in the absence of disease progression or unacceptable toxicity. Beginning in cycle 2, patients receive nivolumab IV over 30 minutes on day 1, etoposide IV on days 1-3, ifosfamide IV continuously over 24 hours on day 2, and carboplatin IV on day 2. Treatment repeats every 21 days for up to 3 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically documented or cytologically confirmed Hodgkin lymphoma; confirmation must include CD30 expression
* Patients must be either refractory to or relapsed after only induction therapy; patients who do not achieve CR after induction therapy are considered primary refractory and are allowed to enter study
* > 40 kg
* Absolute neutrophil count (ANC) >= 1500/uL; filgrastim can be given before and during treatment to achieve target ANC >= 1500 uL
* Platelet (Plt) >= 75,000/uL
* Hemoglobin >= 8.5 g/dl
* Platelet transfusion and packed red blood cell transfusion can also be given prior to the start of treatment and treatment to achieve a target plt >= 75,000/uL and hemoglobin of >= 8.5 g/dl, provided that patients have not received growth factors for at least 14 days prior to entering trial
* Patients must have measurable disease > 1.5 cm evidenced by computed tomography (CT) scan of the neck/chest/abdomen/pelvis or CT/positron emission tomography (PET) scans
* Life expectancy of greater than 3 months
* Eastern Cooperative Oncology Group (ECOG) of 0-2
* Documented informed consent/assent of the participant or legally responsible guardian
* Diffusion capacity of the lung for carbon monoxide (DLCO) >= 60%
* Total bilirubin with 1.5 x the upper limit of normal (ULN) institutional limits; patients with elevation of unconjugated bilirubin alone, as in Gilbert's disease, are eligible
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 3.0 x the institutional upper limit of normal (unless demonstrated Hodgkin lymphoma involvement of the liver); estimated creatinine clearance >= 30 ml/min (Cockcroft-Gault) and/or 24 urine analysis as needed
* For patients with Hodgkin lymphoma (HL) involvement of the liver, AST/ALT < 5.0 x institutional ULN; total bilirubin within 3.0 x institutional ULN; (although patients with HL involvement of the liver are frequently excluded from trials, their liver function tests often improve after treatment; the studies that led to nivolumab approval did not reveal any increased signals of liver toxicities attributed to nivolumab)
* Prothrombin time (PT)/international normalized ration (INR) < 1.5 x ULN and partial thromboplastin time (PTT) (activated [a]PTT) < 1.5 x ULN
* Female subject is either post-menopausal, surgically sterilized, or willing to use and acceptable method of birth control (i.e., a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study; women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of nivolumab
* Men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year; men receiving nivolumab and who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 31 weeks after the last dose of investigational product; women who are not of childbearing potential (i.e., who are postmenopausal or surgically sterile) as well as azoospermic men do not require contraception
* All participants will undergo standard written informed consent procedures as dictated by the City of Hope Human Research Protections Office prior to performing any screening procedures that are not part of standard-of-care; informed consent will be obtained by the principal investigator, collaborating investigators, or other Institutional Review Board (IRB) designated personnel who will meet the training requirements established by the IRB; with the support of research personnel, he/she will explain the nature, duration, purpose of the study, potential risks, alternatives and potential benefits, and all other information contained in the informed consent document; in addition, they will review the experimental subject's bill of rights and the Health Insurance Portability and Accountability Act (HIPAA) research authorization form; prospective research participants will be informed that they may withdraw from the study at any time and for any reason without prejudice; prospective research participants will be afforded sufficient time to consider whether or not to participate in the research
* Patient must be either refractory to or relapsed after 1 line of therapy; prior radiation therapy is allowed
* INCLUSION CRITERIA FOR COHORT B:
* B symptoms at relapse
* Extranodal disease at relapse
* Primary refractory disease
* Relapsed < 1 year after completion of frontline therapy
* Have received brentuximab vedotin as initial therapy

Exclusion Criteria:

* Prior exposure to PD-1 or PD-L1 inhibitors is not allowed
* Must not have had second line chemotherapy for Hodgkin lymphoma
* Active autoimmune diseases requiring systemic treatments
* Vaccinated with live, attenuated vaccine within 4 weeks of first dose of study drug
* Any life-threatening illness, medical condition, or organ system dysfunction that, in the investigator's opinion, could compromise the subject's safety or put the study outcomes at undue risk
* Unwilling or unable to participate in all required study evaluations and procedures
* Unable to understand the purpose and risks of the study and to provide a signed and dated informed consent for (ICF) and authorization to use protected health information (in accordance with national and local subject privacy regulations)
* Patients should not have any uncontrolled illness including ongoing or active infection
* Patients may not be receiving any other investigational agents, or concurrent biological therapy, chemotherapy, or radiation therapy
* Patients must not have received prior chemotherapy or radiation for =< 3 weeks before study enrollment, or those who have not recovered from the adverse events due to agents administered more than 3 weeks earlier are excluded
* Myocardial infarction within 6 months prior to enrollment or New York Heart Association (NYHA) class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities; prior study entry, any electrocardiogram (ECG) abnormality at screening has to be documented by the investigator as not medically relevant
* Significant screening electrocardiogram (ECG) abnormalities including, but not limited to, left bundle branch block, 2nd degree atrioventricular (AV) block type II, 3rd degree block, or corrected QT interval (QTc) >= 470 msec; subjects with a cardiac pacemaker who have a QTc interval of >= 470 msec may be eligible if these findings are considered not clinically significant as documented via a cardiology evaluation
* DLCO < 60%; the clinical studies in support of accelerated approval for nivolumab in chronic (c)HL after failure of ASCT required DLCO > 60%; certain HL induction regimens have the potential for pulmonary toxicity, and nivolumab carries the potential of pneumonitis or other pulmonary toxicities
* Diagnosed or treated for another malignancy within 3 years of enrollment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy, or low-risk prostate cancer after curative therapy
* Patients with active central nervous system (CNS) disease or history of brain metastases are excluded from study
* Patients should be excluded if they have a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration; inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease
* Pregnant women are excluded from this study because of the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk of adverse events in nursing infants secondary to treatment of the mother, breastfeeding should be discontinued
* Recent infection requiring systemic treatment that was completed =< 14 days before the first dose of study drug
* Known history of human immunodeficiency virus (HIV), hepatitis C virus (HCV) or hepatitis B virus (HBV) infection; subjects who are positive for hepatitis B core antibody or hepatitis B surface antigen must have a negative polymerase chain reaction (PCR) result before enrollment, those who are PCR positive will be excluded; subjects who have an undetectable HIV viral load with CD4 >= 300 and are on highly active antiretroviral therapy (HAART) medication are allowed; previously treated hepatitis C patients are also allowed; as there is potential for hepatic toxicity with nivolumab or nivolumab/ipilimumab combinations, drugs with a predisposition to hepatoxicity should be used with caution in patients treated with nivolumab-containing regimen
* History of allergy or adverse drug reaction to study components

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2017-04-24 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2026-04-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Alex F Herrera, Principal Investigator — City of Hope Medical Center
Locations (4):
- United States (4):
  - City of Hope Medical Center, Duarte, California
  - Yale University, New Haven, Connecticut
  - M D Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

REFERENCES:
- [Derived] Mei MG, Lee HJ, Palmer JM, Chen R, Tsai NC, Chen L, McBride K, Smith DL, Melgar I, Song JY, Bonjoc KJ, Armenian S, Nwangwu M, Lee PP, Zain J, Nikolaenko L, Popplewell L, Nademanee A, Chaudhry A, Rosen S, Kwak L, Forman SJ, Herrera AF. Response-adapted anti-PD-1-based salvage therapy for Hodgkin lymphoma with nivolumab alone or in combination with ICE. Blood. 2022 Jun 23;139(25):3605-3616. doi: 10.1182/blood.2022015423. PMID 35316328

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort A (Nivolumab, Etoposide, Ifosfamide, Carboplatin) | Cohort B (Nivolumab, Etoposide, Ifosfamide, Carboplatin)
Started | 43 | 35
Completed | 43 | 35
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A (Nivolumab, Etoposide, Ifosfamide, Carboplatin) | Cohort B (Nivolumab, Etoposide, Ifosfamide, Carboplatin) | Total
Number analyzed (Participants) | 43 | 35 | 78
Age, Continuous [Median (Full Range); unit: years] | 35 [18 to 70] | 30 [19 to 70] | 31.5 [18 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 14 | 31
  Male | 26 | 21 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 11 | 19
  Not Hispanic or Latino | 34 | 24 | 58
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 5 | 2 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 33 | 29 | 62
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 43 | 35 | 78
Bulky Disease at Baseline [Count of Participants; unit: Participants] | 8 | 4 | 12
B Symptoms at Baseline [Count of Participants; unit: Participants] | 15 | 6 | 21
Extranodal Disease at Baseline [Count of Participants; unit: Participants] | 16 | 10 | 26

OUTCOME MEASURES:

1. Primary Outcome: Complete Response Rate by Lugano Classification
Description: Complete response rates were calculated as the percent of evaluable patients that have confirmed complete response by radiographic response including computed tomography and/or positron emission tomography scans; 95% Clopper Pearson confidence limits were calculated for this estimate.
Time Frame: From the initial treatment to the end of the treatment, up to 6 months.
Population: 1 participant in Cohort A and 3 participants in Cohort B were not evaluable for treatment response.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A (Nivolumab, Etoposide, Ifosfamide, Carboplatin) | Cohort B (Nivolumab, Etoposide, Ifosfamide, Carboplatin)
Number analyzed (Participants) | 42 | 32
percentage of participants | 71 [55 to 84] | 88 [71 to 96]

2. Primary Outcome: Number of Participants With Unacceptable Adverse Events
Description: Toxicities were assessed and reported using the Bearman (non-hematologic) and National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 scales. Unacceptable toxicity in a given patient is defined as any non-hematologic or hematological grade 3/4 toxicity that did not resolve to a grade 1/2 within 14 days per NCI CTCAE v4.03 toxicity criteria and was considered at least possibly related to nivolumab and/or ICE, or any other regimen-related cause of death.
Time Frame: From initial treatment to the end of the study, up to 77 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A (Nivolumab, Etoposide, Ifosfamide, Carboplatin) | Cohort B (Nivolumab, Etoposide, Ifosfamide, Carboplatin)
Number analyzed (Participants) | 43 | 35
Participants | 0 | 0

3. Secondary Outcome: Overall Response Rate
Description: Overall response rate was calculated as the percent of evaluable patients that have confirmed complete response or partial remission by radiographic response including computed tomography and/or positron emission tomography scans; 95% Clopper Pearson confidence limits were calculated for this estimate.
Time Frame: From the initial treatment to the end of the treatment, up to 6 months.
Population: 1 participant in Cohort A and 3 participants in Cohort B were not evaluable for treatment response.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A (Nivolumab, Etoposide, Ifosfamide, Carboplatin) | Cohort B (Nivolumab, Etoposide, Ifosfamide, Carboplatin)
Number analyzed (Participants) | 42 | 32
percentage of participants | 81 [66 to 91] | 100 [89 to 100]

4. Secondary Outcome: Two-Year Overall Survival (OS) Rate
Description: Overall survival (OS) is defined as the duration of time from start of study treatment to time of death (due to any cause). OS rate was estimated using the product-limit method of Kaplan and Meier. The event is death.
Time Frame: 2 years from start of treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A (Nivolumab, Etoposide, Ifosfamide, Carboplatin) | Cohort B (Nivolumab, Etoposide, Ifosfamide, Carboplatin)
Number analyzed (Participants) | 43 | 35
percentage of participants | 95 [82 to 99] | 100 [100 to 100]

5. Secondary Outcome: Two-Year Progression-Free Survival (PFS) Rate
Description: Progression-free survival is defined as the duration of time from start of study treatment to time of progression or death, whichever occurs first. PFS rate was estimated using the product-limit method of Kaplan and Meier. The event is progression/relapse or death.
Time Frame: 2 years from start of treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A (Nivolumab, Etoposide, Ifosfamide, Carboplatin) | Cohort B (Nivolumab, Etoposide, Ifosfamide, Carboplatin)
Number analyzed (Participants) | 43 | 35
percentage of participants | 72 [56 to 83] | 94 [77 to 98]

6. Secondary Outcome: Two-Year Progression-Free Survival Rate (Post Autologous Transplant)
Description: Progression-free survival (PFS) is defined as the duration of time from start of transplant to time of progression or death, whichever occurs first. PFS rate was estimated using the product-limit method of Kaplan and Meier. The event is post-transplant progression/relapse or death.
Time Frame: From start of transplant to time of progression, death (due to any cause), or last contact, whichever comes first, assessed 2 years post-transplant, up to 3 years.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A (Nivolumab, Etoposide, Ifosfamide, Carboplatin) | Cohort B (Nivolumab, Etoposide, Ifosfamide, Carboplatin)
Number analyzed (Participants) | 33 | 32
percentage of participants | 94 [77 to 98] | 97 [80 to 100]

7. Secondary Outcome: Cumulative Incidence of Relapse/Progression at 2 Years
Description: The cumulative incidence of relapse/progression was calculated as competing risks using the method of Gooley et al. The event is relapse/progression. Deaths without relapse/progression are considered a competing risk.
Time Frame: 2 years from start of treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A (Nivolumab, Etoposide, Ifosfamide, Carboplatin) | Cohort B (Nivolumab, Etoposide, Ifosfamide, Carboplatin)
Number analyzed (Participants) | 43 | 35
percentage of participants | 9 [4 to 24] | 6 [2 to 24]

8. Secondary Outcome: Non-relapse Mortality (NRM) at 2 Years
Description: The cumulative incidence of non-relapse mortality was calculated as competing risks using the method of Gooley et al. NRM is defined as death occurring in a patient from causes other than relapse or progression. Deaths from relapse/progression are considered a competing risk.
Time Frame: 2 years from start of treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A (Nivolumab, Etoposide, Ifosfamide, Carboplatin) | Cohort B (Nivolumab, Etoposide, Ifosfamide, Carboplatin)
Number analyzed (Participants) | 43 | 35
percentage of participants | 2 [0.3 to 16] | 0 [0 to 0]

ADVERSE EVENTS:
Time Frame: Adverse events and all-cause mortality were monitored/assessed from initial treatment to the end of protocol follow-up, up to 77 months.
Arm/Group | Cohort A (Nivolumab, Etoposide, Ifosfamide, Carboplatin) | Cohort B (Nivolumab, Etoposide, Ifosfamide, Carboplatin)
All-Cause Mortality (participants affected / at risk) | 2/43 | 0/35
Serious Adverse Events (participants affected / at risk) | 5/43 | 3/35
Other Adverse Events (participants affected / at risk) | 42/43 | 34/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A (Nivolumab, Etoposide, Ifosfamide, Carboplatin) (N=43) | Cohort B (Nivolumab, Etoposide, Ifosfamide, Carboplatin) (N=35)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0)
Thyroiditis (Endocrine disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 0 (0) | 2 (2)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Altered Mental Status (Nervous system disorders) | 1 (1) | 0 (0)
Unintended pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Renal Failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Aspiration, Intubation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A (Nivolumab, Etoposide, Ifosfamide, Carboplatin) (N=43) | Cohort B (Nivolumab, Etoposide, Ifosfamide, Carboplatin) (N=35)
ANEMIA (Blood and lymphatic system disorders) | 12 (23) | 27 (42)
PALPITATIONS (Cardiac disorders) | 0 (0) | 2 (2)
SINUS BRADYCARDIA (Cardiac disorders) | 1 (1) | 3 (5)
SINUS TACHYCARDIA (Cardiac disorders) | 7 (7) | 19 (30)
EAR PAIN (Ear and labyrinth disorders) | 1 (2) | 0 (0)
VERTIGO (Ear and labyrinth disorders) | 0 (0) | 1 (1)
HYPERTHYROIDISM (Endocrine disorders) | 2 (5) | 3 (3)
HYPOTHYROIDISM (Endocrine disorders) | 0 (0) | 1 (1)
BLURRED VISION (Eye disorders) | 3 (5) | 2 (3)
CONJUNCTIVITIS (Eye disorders) | 1 (1) | 0 (0)
DRY EYE (Eye disorders) | 0 (0) | 1 (1)
SWELLING EYE (Eye disorders) | 1 (1) | 0 (0)
VISUAL DISTURBANCE (Eye disorders) | 1 (1) | 0 (0)
VITREOUS HEMORRHAGE (Eye disorders) | 1 (1) | 0 (0)
WATERING EYES (Eye disorders) | 1 (1) | 1 (1)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 1 (1) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 6 (8) | 4 (5)
BLOATING (Gastrointestinal disorders) | 2 (3) | 0 (0)
BLOOD IN STOOL (Gastrointestinal disorders) | 0 (0) | 1 (1)
BLOODY STOOL (Gastrointestinal disorders) | 0 (0) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 8 (10) | 14 (15)
DIARRHEA (Gastrointestinal disorders) | 6 (10) | 4 (4)
DRY MOUTH (Gastrointestinal disorders) | 0 (0) | 1 (2)
DYSPEPSIA (Gastrointestinal disorders) | 2 (2) | 0 (0)
FLATULENCE (Gastrointestinal disorders) | 2 (2) | 0 (0)
GERD SYMPTOMS (Gastrointestinal disorders) | 0 (0) | 1 (1)
HEARTBURN (Gastrointestinal disorders) | 0 (0) | 1 (1)
LIP PAIN (Gastrointestinal disorders) | 1 (1) | 0 (0)
MUCOSITIS ORAL (Gastrointestinal disorders) | 3 (6) | 2 (3)
NAUSEA (Gastrointestinal disorders) | 15 (22) | 26 (41)
STOMACH DISCOMFORT (Gastrointestinal disorders) | 1 (1) | 0 (0)
TOOTHACHE (Gastrointestinal disorders) | 2 (2) | 1 (1)
VOMITING (Gastrointestinal disorders) | 8 (9) | 16 (21)
CHILLS (General disorders) | 5 (6) | 4 (4)
EDEMA FACE (General disorders) | 0 (0) | 2 (2)
EDEMA HANDS (General disorders) | 1 (1) | 0 (0)
EDEMA LIMBS (General disorders) | 2 (3) | 2 (2)
FATIGUE (General disorders) | 19 (33) | 24 (34)
FEET (General disorders) | 1 (1) | 0 (0)
FEVER (General disorders) | 8 (12) | 3 (3)
GLUCOSURIA (General disorders) | 0 (0) | 1 (1)
INFUSION RELATED REACTION (General disorders) | 3 (3) | 0 (0)
INJECTION SITE REACTION (General disorders) | 0 (0) | 2 (2)
MALAISE (General disorders) | 1 (1) | 0 (0)
NECK EDEMA (General disorders) | 1 (1) | 0 (0)
NON-CARDIAC CHEST PAIN (General disorders) | 2 (2) | 3 (3)
PAIN (General disorders) | 3 (5) | 1 (1)
RUNNY NOSE (General disorders) | 0 (0) | 1 (1)
SCALP SENSITIVITY (General disorders) | 0 (0) | 1 (1)
ALLERGIC REACTION (Immune system disorders) | 0 (0) | 2 (2)
COVID-19 (Infections and infestations) | 0 (0) | 2 (2)
PAPULOPUSTULAR RASH (Infections and infestations) | 0 (0) | 1 (1)
PARONYCHIA (Infections and infestations) | 0 (0) | 1 (1)
PERIANAL FOLLICULITS (Infections and infestations) | 0 (0) | 1 (1)
PICC LINE ISSUES (Infections and infestations) | 1 (1) | 0 (0)
RASH PUSTULAR (Infections and infestations) | 1 (2) | 0 (0)
SEPSIS (Infections and infestations) | 1 (1) | 0 (0)
TOOTH INFECTION (Infections and infestations) | 1 (1) | 0 (0)
UPPER RESPIRATORY INFECTION (Infections and infestations) | 3 (3) | 0 (0)
VAGINAL INFECTION (Infections and infestations) | 3 (3) | 0 (0)
YEAST INFECTION (Infections and infestations) | 1 (1) | 0 (0)
ACTIVATED PARTIAL THROMBOPLASTIN TIME PROLONGED (Investigations) | 3 (9) | 5 (6)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 11 (17) | 8 (8)
ALKALINE PHOSPHATASE INCREASED (Investigations) | 5 (10) | 3 (3)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 7 (10) | 4 (4)
BLOOD BILIRUBIN INCREASED (Investigations) | 4 (5) | 0 (0)
CREATININE INCREASED (Investigations) | 3 (4) | 0 (0)
EOSINOPHILIA (Investigations) | 1 (2) | 0 (0)
HEMOGLOBIN INCREASED (Investigations) | 1 (1) | 0 (0)
LYMPHOCYTE COUNT DECREASED (Investigations) | 4 (7) | 8 (13)
NEUTROPHIL COUNT DECREASED (Investigations) | 9 (14) | 12 (15)
PLATELET COUNT DECREASED (Investigations) | 8 (23) | 11 (20)
WEIGHT GAIN (Investigations) | 2 (2) | 5 (9)
WEIGHT LOSS (Investigations) | 3 (3) | 2 (2)
WHITE BLOOD CELL DECREASED (Investigations) | 9 (17) | 11 (15)
ACIDOSIS (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
ALKALOSIS (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
ANOREXIA (Metabolism and nutrition disorders) | 2 (2) | 9 (9)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
HYPERCALCEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 6 (8) | 1 (2)
HYPERKALEMIA (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
HYPERURICEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPOALBUMINEMIA (Metabolism and nutrition disorders) | 4 (7) | 1 (1)
HYPOCALCEMIA (Metabolism and nutrition disorders) | 4 (4) | 2 (2)
HYPOGLYCEMIA (Metabolism and nutrition disorders) | 7 (16) | 3 (4)
HYPOKALEMIA (Metabolism and nutrition disorders) | 7 (12) | 4 (5)
HYPOMAGNESEMIA (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
HYPONATREMIA (Metabolism and nutrition disorders) | 11 (13) | 4 (7)
HYPOPHOSPHATEMIA (Metabolism and nutrition disorders) | 6 (10) | 2 (2)
OBESITY (Metabolism and nutrition disorders) | 1 (1) | 3 (4)
TUMOR LYSIS SYNDROME (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 7 (10) | 4 (5)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 9 (14) | 5 (5)
BILATERAL KNEE PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
CRAMPING (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
GENERALIZED MUSCLE WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
MUSCLE WEAKNESS LOWER LIMB (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MYALGIA (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
PERIRECTAL LUMP/ BULGE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
AMNESIA (Nervous system disorders) | 1 (1) | 0 (0)
DIZZINESS (Nervous system disorders) | 3 (3) | 1 (1)
DYSGEUSIA (Nervous system disorders) | 0 (0) | 5 (5)
HEADACHE (Nervous system disorders) | 9 (9) | 7 (7)
HYPERSOMNIA (Nervous system disorders) | 0 (0) | 1 (1)
LETHARGY (Nervous system disorders) | 1 (1) | 0 (0)
NEUROPATHIC PAIN (Nervous system disorders) | 1 (1) | 0 (0)
PARESTHESIA (Nervous system disorders) | 1 (1) | 0 (0)
PERIPHERAL MOTOR NEUROPATHY (Nervous system disorders) | 1 (4) | 0 (0)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 4 (4) | 5 (5)
SOMNOLENCE (Nervous system disorders) | 1 (1) | 0 (0)
SYNCOPE (Nervous system disorders) | 1 (1) | 0 (0)
AGITATION (Psychiatric disorders) | 1 (1) | 1 (2)
ANXIETY (Psychiatric disorders) | 7 (9) | 6 (6)
DEPRESSION (Psychiatric disorders) | 2 (2) | 0 (0)
INSOMNIA (Psychiatric disorders) | 4 (4) | 5 (6)
RESTLESSNESS (Psychiatric disorders) | 1 (1) | 0 (0)
BACTERIA 2+ ON UA (Renal and urinary disorders) | 0 (0) | 1 (1)
BLADDER PRESSURE (Renal and urinary disorders) | 0 (0) | 2 (2)
CHRONIC KIDNEY DISEASE (Renal and urinary disorders) | 1 (1) | 0 (0)
DYSURIA (Renal and urinary disorders) | 1 (1) | 9 (11)
HEMATURIA (Renal and urinary disorders) | 0 (0) | 6 (6)
HEMORRHAGIC CYSTITIS (Renal and urinary disorders) | 0 (0) | 2 (2)
PROTEINURIA (Renal and urinary disorders) | 0 (0) | 5 (5)
URINARY FREQUENCY (Renal and urinary disorders) | 1 (2) | 3 (3)
URINARY TRACT PAIN (Renal and urinary disorders) | 0 (0) | 2 (2)
BREAST PAIN (Reproductive system and breast disorders) | 0 (0) | 1 (1)
MENORRHAGIA (Reproductive system and breast disorders) | 1 (4) | 0 (0)
PELVIC PAIN (Reproductive system and breast disorders) | 0 (0) | 1 (1)
VAGINAL PAIN (Reproductive system and breast disorders) | 0 (0) | 1 (1)
ALLERGIC RHINITIS (Respiratory, thoracic and mediastinal disorders) | 4 (8) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 3 (3)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 7 (8)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (3)
HOARSENESS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 2 (2)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
POSTNASAL DRIP (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
SORE THROAT (Respiratory, thoracic and mediastinal disorders) | 3 (7) | 0 (0)
ALOPECIA (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
BULLOUS DERMATITIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
CYSTIC LESION (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
DRY SKIN (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
HYPOHIDROSIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
PALLOR (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
PRURITUS (Skin and subcutaneous tissue disorders) | 10 (10) | 6 (8)
RASH ACNEIFORM (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 13 (16) | 3 (4)
WART (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 (0) | 1 (1)
FLUSHING (Vascular disorders) | 1 (2) | 1 (1)
HOT FLASHES (Vascular disorders) | 1 (1) | 3 (4)
HYPERTENSION (Vascular disorders) | 12 (25) | 20 (40)
HYPOTENSION (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-27): https://cdn.clinicaltrials.gov/large-docs/71/NCT03016871/Prot_SAP_000.pdf